CLINICAL TRIAL: NCT04586192
Title: Developing and Assessing a Digital Mental Health and Wellness Intervention for Adults: Randomized Control Trial of the Common Elements Toolbox (COMET)
Brief Title: Digital Mental Health and Wellness Intervention for Adults: A Randomized Control Trial of COMET
Acronym: COMET
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 30845924
Record Dates: First submitted 2020-10-05; First posted 2020-10-14 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-10

CONDITIONS: Depressive Symptoms; Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- COMET (Experimental): Participants receive modules focused on cognitive restructuring, gratitude, behavioral activation and self-compassion. Participants were randomized to receive 3 of the 4 possible modules: behavioral activation, cognitive restructuring, gratitude, and self-compassion.Participants in the intervention condition were randomized to receive descriptions of the four modules at the beginning of the intervention that were phrased to focus on building and improving strengths (positive) or reducing negative emotions and behaviors (negative).
  Interventions: Other: Common Elements Toolbox- Adult version (COMET-A)
- Self-Awareness Control (Sham Comparator): Participants learn about self-awareness through writing about memories, writing a short argumentative essay, and noticing objects in their surroundings.
  Interventions: Other: Self-awareness Control
- Waitlist (No Intervention): Participants filled out all pre-test and post-test measures without having access to COMET of the active control exercises. Participants in this condition will receive access to COMET at the end of the study.

INTERVENTIONS:
Other: Common Elements Toolbox- Adult version (COMET-A) — COMET includes four different modules that teach participants exercises designed to improve mental health and well-being. Participants are asked to complete exercises focused on behavioral activation, cognitive restructuring, gratitude and self-compassion. At the end of the intervention, participants are sent templates that they can you to complete the exercises on, and are encouraged to continue practicing their exercises in their daily life.
  Arms: COMET
Other: Self-awareness Control — A control condition in which participants learn about self-awareness through writing about memories, writing a short argumentative essay, and noticing objects in their surroundings.
  Arms: Self-Awareness Control

SUMMARY:
The investigators are evaluating the acceptability and effectiveness of brief online wellness modules. Participants will be randomly assigned to the intervention condition, an active control condition, or a wait-list control condition. The investigators are using a factorial design, such that each participant in the intervention condition will be randomly assigned to receive three of four wellness modules.

The investigators will analyze the intervention's effectiveness as a universal intervention (using the full sample) and a targeted intervention (using the subset of the sample that reported elevated depressive symptoms or anxiety symptoms at baseline).

ELIGIBILITY:
Adult participants (at least 18 years old) will be eligible for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2500 (Estimated)
Dates: Start 2021-01-31 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in Patient Health Questionnaire-9 (PHQ-9) | Up to 12 weeks post-intervention
  Depression questionnaire. Scores range from 0 to 27. Lower scores indicate less depression.
Change in Generalized Anxiety Disorder Screener-7 (GAD-7) | Up to 12 weeks post-intervention
  Anxiety questionnaire. Total scores range from 0-21. Lower scores indicate less anxiety.
Change in Short Warwick-Edinburgh Mental Well-being Scale (SWEMWBS) | Up to 12 weeks post-intervention
  Subjective Well-being questionnaire. Total scores range from 7 to 35. Higher values indicate higher well-being scores.
Ratings of Acceptability of Intervention Measure (AIM) | Immediately after the intervention
  Questionnaire measuring the acceptability of an intervention. Acceptability refers to the perception that a given treatment is agreeable or satisfactory. The total score ranges from 4 to 20. Higher scores indicate higher acceptability ratings.
Mechanism Questions | Up to 12 weeks post-intervention
  Participants answered questions relating to each module's mechanism of change on a 7-point Likert Scale, from "strongly disagree" to "strongly agree".
  Specifically, we asked participants:
  * How capable they feel about managing negative thoughts
  * If they will intentionally spend time doing activities they enjoy
  * If they will notice and appreciate good things
  * If they will be able to treat themselves with empathy and compassion
Ability to Cope with COVID-19 | Up to 12 weeks post-intervention
  2 questions related to their ability to cope with stressors over the upcoming weeks (including challenges relating to COVID-19). Participants answered these questions on a 7-point Likert Scale, from "strongly disagree" to "strongly agree". Specifically, we asked participants:
  * if they will be able to handle lifestyle changes due to the coronavirus,
  * if the pandemic will have an extremely negative impact on their life.
Secondary Control | Up to 12 weeks post-intervention
  We asked participants three items to assess secondary control (Weisz et al., 2010). The items are scored on a 4-point Likert scale, ranging from 0 ("Very false") to 3 ("Very true").
  The three items are:
  * When something bad happens, I can find a way to think about it that makes me feel better.
  * After a really hard day, I can make myself feel better by remembering some good things that happened.
  * When bad things happen to me that I can't control, there are lots of things I can do to feel better.
  Higher scores will indicate greater secondary control.
Perceived Utility | Immediately after the intervention
  Participants were asked to rate three items relating to the perceived utility of each module. Specifically, we asked participants:
  * How helpful the module was
  * How engaging the module was
  * How much they will continue applying content from the module
  Higher scores will indicate greater perceived utility.

CONTACTS AND LOCATIONS:
Overall Officials: Robert J DeRubeis, PhD, Study Director — University of Pennsylvania; Akash Wasil, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No